CLINICAL TRIAL: NCT03065998
Title: Double Blind Placebo Control Opipramol-Baclofen Treatment for Addiction: Medical and Cognitive Effects
Brief Title: Double Blind Placebo Control Opipramol-Baclofen Treatment for Addiction
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Israel (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 066-2017 MOH
Record Dates: First submitted 2017-02-14; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Opipramol; Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-A (Active Comparator): opripramol 150 mg per day (3*50) Opipramol is a selective agonist for sigma-1 receptor. It is clinically used as an antidepressant and anxiolytic agent.
  Interventions: Drug: Opipramol; Drug: Baclofen
- Drug-B (Active Comparator): baclofen 90 mg per day (3*30) Baclofen is a GABAb-1 antagonist and has shown partial efficacy in suppressing withdrawal symptoms in alcohol addicts and cocaine.
  Interventions: Drug: Opipramol; Drug: Baclofen

INTERVENTIONS:
Drug: Opipramol — PO
Drug: Baclofen — PO

SUMMARY:
The aim of this study is examining the combination of two FDA approved drugs, Opipramol and baclofen, which may increase rehabilitation from psychoactive substances. Previous studies have indicated a connection of sigma-1 receptor to cocaine abuse and raised the possibility that these receptors as mediators of drug craving . However previous studies showed partial efficacy with no significant relapse in relapse rates. The same is true for the use of GABAb-1 receptor antagonist. Opipramol is a selective agonist for sigma-1 receptor. It is clinically used as an antidepressant and anxiolytic agent. Moreover, previous open and controlled trials indicated that the GABAb-1 antagonist baclofen partial efficacy in suppressing withdrawal symptoms in alcohol addicts and cocaine. Our studies in an animal model for addiction have shown a significant effect of the combine treatment of the indicated medications both in decreasing relapse and increase of -number of respondents.

ELIGIBILITY:
Inclusion Criteria:

* Age will be 60-18, both sexes, seeking treatment in order to stop the consumption of materials

Exclusion Criteria:

* Did not include trial addicts with co-morbidity, kidney, heart, metabolic, neurological and psychiatric disorders (psychosis, chronic depression).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Decreased craving | 1 month
  Lower withdrawal symptom will be measured by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Gal Yadid, PhD, Principal Investigator — Bar Ilan University
Locations (1):
- Retorno rehabilitation center, Bet Shemesh, Israel

IPD SHARING:
Plan to Share IPD: Undecided